CLINICAL TRIAL: NCT02658500
Title: Short and Long Term Effect of Early Infant Feeding and Nutritional Status on the Children's Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Sanyuan Foods Co Ltd (Industry)
Collaborators: Capital Institute of Pediatrics, China (Other); Peking University (Other); Beijing Ditan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: D14110000481400
Record Dates: First submitted 2016-01-14; First posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Health Behavior
Keywords: early infant feeding; infant intestinal flora; infant health
MeSH Terms: conditions — Health Behavior | interventions — Infant Formula; Milk, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infant Formula (Experimental): 200 newborns just consume the infant formula from 0-42 days to six months age.
  Interventions: Dietary Supplement: Infant Formula
- Breast Milk (Other): 100 newborns were just fed with breast milk from after birth to six months age.
  Interventions: Dietary Supplement: breast milk

INTERVENTIONS:
Dietary Supplement: Infant Formula
  Other Names: superior quality infant formula
  Arms: Infant Formula
Dietary Supplement: breast milk
  Arms: Breast Milk

SUMMARY:
This study evaluates the early infant feeding in the infant intestinal microecology and the long term health. 300 healthy term newborns were involved into the study on its first stage. Depending on the type of feeding the infants were divided into 3 groups with random allocation to one of the formula feeding groups: the group A included 100 infants consuming the formula supplement with superior quality whey protein, the group B -100 infants fed with a standard formula, and the group C -100 infants who were breastfed.

DETAILED DESCRIPTION:
Throughout the human lifetime, the intestinal microbiota performs vital functions, such as barrier function, metabolic reactions, trophic effects, and maturation of the host's innate and adaptive immune responses. Therefore, the human health depends on the gut health. It is reported that the human gut microbiota of a healthy adult is highly resilient and very stable over time. And before it reaches maturity, the microbiota must develop itself from birth and establish its mutually beneficial cohabitation with the host. However, the early developments of the microbiota in infants are influenced by many factors, such as prenatal parameters, the influence of the mother and her microbiota, and therapies occurring around the time of birth.

Human milk is the sole source of nutrition for infants during the first weeks to months after birth, and has evolved to provide nutrition and immunological protection in the extra-uterine environment into which the infant is born. But when breastfeeding is not possible, human newborns may circumstantially be fed with infant formulas. The difference of feeding mode has been demonstrated to have a strong influence on early gut colonization particularly on the probiotic bacteria. Studies show that breastfed infants have higher counts of Bifidobacteria and Lactobacillus and lower counts of Bacteroides, Clostridium, coccoides group, Staphylococcus, and Enterobacteriaceae as compared with formula-fed infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term newborns (the mean gestational age in weeks > 36.0) with birth weight ≥2500 g appropriate for gestational age
* Apgar scores > 7
* Uncomplicated early course of neonatal period
* Impossibility of breastfeeding (for infants randomized into the bottle-feeding groups)

Exclusion Criteria:

* The minimum possibility of breastfeeding (for infants randomized into the bottle-feeding groups)
* The diagnosis of a significant chronic medical condition including: HIV infection; cancer; bone marrow or organ transplantation; blood product administration within the last 3 mo; bleeding disorder; known congenital malformation or genetic disorder
* If the parent or legal guardian were unable to read and/or comprehend Chinese
* If the family moved outside of Beijing during the study period (i.e., would be unavailable for follow-up)

Max Age: 42 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of the compositions of the intestinal microbiota of infants fed formula and breast milk by high-throughput sequencing | up to 8 months
  At the age of 1, 2, 3, 6 months, 2 g fecal samples were collected from diapers after defaecation, immediately put into a sterile plastic containers and stored at -20℃ until they were transported (within 24 hours) to the technology center of Beijing Sanyuan Foods Co. Then, each sample was frozen at -80℃ until further processing. The samples were transported on dry ice.
  The analysis methods of fecal samples include high-throughput gene sequencing and quantitative real-time PCR for analysis of Bifidobacterium, Lactobacillus, escherichia coli and Candida fungi etc.

CONTACTS AND LOCATIONS:
Overall Officials: CHEN LIJUN, Study Director — Beijing Sanyuan Foods Co Ltd
Locations (4):
- China (4):
  - Beijing Ditan Hospital Capital Mendical University, Beijing, Beijing Municipality
  - Tongzhou Matemal & Child Health Hospital of Beijing, Beijing, Beijing Municipality
  - Henan University of Science and Technology, Luoyang, Henan
  - Central South University, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matamoros S, Gras-Leguen C, Le Vacon F, Potel G, de La Cochetiere MF. Development of intestinal microbiota in infants and its impact on health. Trends Microbiol. 2013 Apr;21(4):167-73. doi: 10.1016/j.tim.2012.12.001. Epub 2013 Jan 14. PMID 23332725
- [Background] Rouge C, Goldenberg O, Ferraris L, Berger B, Rochat F, Legrand A, Gobel UB, Vodovar M, Voyer M, Roze JC, Darmaun D, Piloquet H, Butel MJ, de La Cochetiere MF. Investigation of the intestinal microbiota in preterm infants using different methods. Anaerobe. 2010 Aug;16(4):362-70. doi: 10.1016/j.anaerobe.2010.06.002. Epub 2010 Jun 9. PMID 20541022
- [Background] Ahrne S, Lonnermark E, Wold AE, Aberg N, Hesselmar B, Saalman R, Strannegard IL, Molin G, Adlerberth I. Lactobacilli in the intestinal microbiota of Swedish infants. Microbes Infect. 2005 Aug-Sep;7(11-12):1256-62. doi: 10.1016/j.micinf.2005.04.011. Epub 2005 Jun 8. PMID 16002310
- [Background] Endo A, Pӓrtty A, Kalliomӓki M, Isolauri E, Salminen S. Long-term monitoring of the human intestinal microbiota from the 2nd week to 13 years of age. Anaerobe. 2014 Aug;28:149-56. doi: 10.1016/j.anaerobe.2014.06.006. Epub 2014 Jun 13. PMID 24933584
- [Background] Bisgaard H, Li N, Bonnelykke K, Chawes BL, Skov T, Paludan-Muller G, Stokholm J, Smith B, Krogfelt KA. Reduced diversity of the intestinal microbiota during infancy is associated with increased risk of allergic disease at school age. J Allergy Clin Immunol. 2011 Sep;128(3):646-52.e1-5. doi: 10.1016/j.jaci.2011.04.060. Epub 2011 Jul 22. PMID 21782228
- [Background] Kapiki A, Costalos C, Oikonomidou C, Triantafyllidou A, Loukatou E, Pertrohilou V. The effect of a fructo-oligosaccharide supplemented formula on gut flora of preterm infants. Early Hum Dev. 2007 May;83(5):335-9. doi: 10.1016/j.earlhumdev.2006.07.003. Epub 2006 Sep 14. PMID 16978805
- [Background] Chrzanowska-Liszewska D, Seliga-Siwecka J, Kornacka MK. The effect of Lactobacillus rhamnosus GG supplemented enteral feeding on the microbiotic flora of preterm infants-double blinded randomized control trial. Early Hum Dev. 2012 Jan;88(1):57-60. doi: 10.1016/j.earlhumdev.2011.07.002. Epub 2011 Nov 4. PMID 22055271
- [Background] Arboleya S, Ang L, Margolles A, Yiyuan L, Dongya Z, Liang X, Solis G, Fernandez N, de Los Reyes-Gavilan CG, Gueimonde M. Deep 16S rRNA metagenomics and quantitative PCR analyses of the premature infant fecal microbiota. Anaerobe. 2012 Jun;18(3):378-80. doi: 10.1016/j.anaerobe.2012.04.013. Epub 2012 May 8. PMID 22579986
- [Background] Schwiertz A, Gruhl B, Lobnitz M, Michel P, Radke M, Blaut M. Development of the intestinal bacterial composition in hospitalized preterm infants in comparison with breast-fed, full-term infants. Pediatr Res. 2003 Sep;54(3):393-9. doi: 10.1203/01.PDR.0000078274.74607.7A. Epub 2003 Jun 4. PMID 12788986
- [Background] Fallani M, Young D, Scott J, Norin E, Amarri S, Adam R, Aguilera M, Khanna S, Gil A, Edwards CA, Dore J; Other Members of the INFABIO Team. Intestinal microbiota of 6-week-old infants across Europe: geographic influence beyond delivery mode, breast-feeding, and antibiotics. J Pediatr Gastroenterol Nutr. 2010 Jul;51(1):77-84. doi: 10.1097/MPG.0b013e3181d1b11e. PMID 20479681
- [Background] Andersen BL, Farrar WB, Golden-Kreutz DM, Glaser R, Emery CF, Crespin TR, Shapiro CL, Carson WE 3rd. Psychological, behavioral, and immune changes after a psychological intervention: a clinical trial. J Clin Oncol. 2004 Sep 1;22(17):3570-80. doi: 10.1200/JCO.2004.06.030. PMID 15337807
- [Background] Meropol SB, Edwards A. Development of the infant intestinal microbiome: A bird's eye view of a complex process. Birth Defects Res C Embryo Today. 2015 Dec;105(4):228-39. doi: 10.1002/bdrc.21114. Epub 2015 Dec 11. PMID 26663826
- [Background] Wernimont S, Northington R, Kullen MJ, Yao M, Bettler J. Effect of an alpha-lactalbumin-enriched infant formula supplemented with oligofructose on fecal microbiota, stool characteristics, and hydration status: a randomized, double-blind, controlled trial. Clin Pediatr (Phila). 2015 Apr;54(4):359-70. doi: 10.1177/0009922814553433. Epub 2014 Oct 8. PMID 25297064
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Medina Vera I, Velasco Hidalgo L, Alonso Ocana MV. Higher versus lower protein intake in formula-fed term infants. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD013758. doi: 10.1002/14651858.CD013758.pub2. PMID 37929831
- [Derived] Qiao W, Chen J, Zhang M, Wang Y, Yang B, Zhao J, Jiang T, Chen L. A cohort study of vitamins contents in human milk from maternal-infant factors. Front Nutr. 2022 Sep 6;9:993066. doi: 10.3389/fnut.2022.993066. eCollection 2022. PMID 36147300
- [Derived] Chen J, Liu Y, Zhao J, Jiang T, Xu T, Liu B, Liu Y, Yang B, Li Y, Zhang X, Hou J, Chen L. Three urban areas of China: a cohort study of maternal-infant factors and HM protein components. Food Funct. 2022 May 10;13(9):5202-5214. doi: 10.1039/d1fo04123a. PMID 35438093
- [Derived] Zhao J, Yi W, Liu B, Dai Y, Jiang T, Chen S, Wang J, Feng B, Qiao W, Liu Y, Zhou H, He J, Hou J, Chen L. MFGM components promote gut Bifidobacterium growth in infant and in vitro. Eur J Nutr. 2022 Feb;61(1):277-288. doi: 10.1007/s00394-021-02638-5. Epub 2021 Jul 29. PMID 34324046